CLINICAL TRIAL: NCT05727293
Title: A Case Report of a Patient With Intellectual Disability and Neurogenic Bladder Complicated With Sepsis
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2022-469-01
Record Dates: First submitted 2022-12-04; First posted 2023-02-14 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2022-09

CONDITIONS: Sepsis Bacterial
Keywords: intellectual disability；Neurogenic bladder；Sepsis ；

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: noting — Non intervention

SUMMARY:
A case report of a patient with intellectual disability and neurogenic bladder complicated with sepsis

DETAILED DESCRIPTION:
To summarize the individual care experience of a patient with neurogenic cystitis with sepsis and mental retardation. The main points of nursing care include: conducting personalized nuring care for early sepsis; carring out care for urinary incontinence and urinary tract infection; bulinding health-management plans with family members; and a full course of psychologic diversion that alleviates negative feelings among patients and family members.

ELIGIBILITY:
Inclusion Criteria:

Dysgnosia Neurogenic bladder Pyohemia

Exclusion Criteria:

Intellectually normal person No urinary infection

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A patient with neurogenic cystitis with sepsis and mental retardation.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-11-06 (Actual)

PRIMARY OUTCOMES:
Lactic acid | During the first 6 days of ICU stay
  "In some pathological conditions, such as respiratory failure or circulatory failure, tissue hypoxia may be induced, and due to this hypoxia, lactic acid in the body may be elevated." Elevated lactic acid in the body can cause lactic acidosis. Checking the blood lactate level may indicate the severity of the underlying disease.The normal range is 0.05mmol/L-1.7mmol/L.
Sequential Organ Failure Assessment | During the first 3 days of ICU stay
  This scale can describe the dysfunction or failure of individual organs in a continuous form, and can evaluate the degree of mild dysfunction to severe failure. It can be used to measure the occurrence and development of single or whole organ dysfunction repeatedly in clinical research, so as to determine the characteristics describing organ dysfunction or failure, which has a closer relationship with sepsis.
Indicators of infection | During the first 6 days of ICU stay
  Hemameba level
C-reaction protein | During the first 6 days of ICU stay
  Indicators of infection

CONTACTS AND LOCATIONS:
Overall Officials: huiying Fuhuiying, Principal Investigator — colleague
Locations (1):
- One Case of Individualized Nursing Plan for Sepsis, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yang PY, Meng NH, Chou EC. Voiding dysfunctions in children with mental retardation. Neurourol Urodyn. 2010 Sep;29(7):1272-5. doi: 10.1002/nau.20824. PMID 19852064
- [Result] Wehrberger C, Madersbacher S, Jungwirth S, Fischer P, Tragl KH. Lower urinary tract symptoms and urinary incontinence in a geriatric cohort - a population-based analysis. BJU Int. 2012 Nov;110(10):1516-21. doi: 10.1111/j.1464-410X.2012.11022.x. Epub 2012 Mar 12. PMID 22409717
- [Result] Dinh A, Hallouin-Bernard MC, Davido B, Lemaignen A, Bouchand F, Duran C, Even A, Denys P, Perrouin-Verbe B, Sotto A, Lavigne JP, Bruyere F, Grall N, Tavernier E, Bernard L. Weekly Sequential Antibioprophylaxis for Recurrent Urinary Tract Infections Among Patients With Neurogenic Bladder: A Randomized Controlled Trial. Clin Infect Dis. 2020 Dec 15;71(12):3128-3135. doi: 10.1093/cid/ciz1207. PMID 31867616
- [Result] von Gontard A, Hussong J, Yang SS, Chase J, Franco I, Wright A. Neurodevelopmental disorders and incontinence in children and adolescents: Attention-deficit/hyperactivity disorder, autism spectrum disorder, and intellectual disability-A consensus document of the International Children's Continence Society. Neurourol Urodyn. 2022 Jan;41(1):102-114. doi: 10.1002/nau.24798. Epub 2021 Sep 29. PMID 34586694